CLINICAL TRIAL: NCT01950000
Title: Efficacy and Safety of Opioid Analgesics as a Preventive Treatment of Procedural Pain Associated With Turning Among Critically Ill Patients Under Mechanical Ventilation. A Controlled Clinical Trial Comparing Placebo and Fentanyl
Brief Title: Treatment of Procedural Pain Associated With Turning in Patients With Mechanical Ventilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRS-FEN-2010-01
Record Dates: First submitted 2013-09-06; First posted 2013-09-25 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Critical Illness; Pain
Keywords: Pain. Analgesia. Prevention
MeSH Terms: conditions — Critical Illness; Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo Treatment: A sterile sodium chloride injection 0.9% 10 ml
  Interventions: Other: Placebo
- Fentanest (Experimental): For this study Fentanest doses were adjusted based on published guidelines from the values recommended media to a whole number and differentiating two groups of patients (multiple trauma / surgical or medical) The maximum dose is 100 mcg Fentanest. The multiple trauma patients / surgical 1.5 mcg / kg and in medical patients 1.0 mcg / kg were given a single bolus Fentanest / Placebo by type of patient (surgical / multiple trauma or physician) 5 'before turning mobilization with personal hygiene.
  The bolus is given slowly (30'') intravenously, to be preferred by a peripheral without vasoactive drugs (only with fluid therapy).
  Pharmaceutical form:
  Sterile solution for injection. Each mL of injectable solution contains the equivalent of 0.05 mg of Fentanest; Excipients: sodium chloride and water for injection.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl
  Arms: Fentanest
Other: Placebo
  Arms: Placebo

SUMMARY:
Background: Few studies have addressed the situation of procedural pain and the use of preemptive analgesia for turning in patients under mechanical ventilation.

Aim: Evaluation effect of preemptive fentanyl on the incidence of pain during turning maneuvers in critically ill patients under mechanical ventilation.

Design: Single-center clinical trial, national, randomized, double-blind, with a parallel group, and two arms of treatment: saline placebo and fentanyl.

Primary Endpoint: Incidence of pain during the turning procedures that are carried out by nurses measured by means of the Behavioral Pain Scale (BPS).

Study Population: Critically ill patients, age > 18 years, admitted to ICU and expected to require mechanical ventilation for at least 24 h.

Sample Size: 80 patients divided into the two groups (40 patients each). Statistical Analysis: A preliminary descriptive analysis will be carried. Later, results of primary end point will be comparing after the eventual corrections of corresponding variables using a multivariable approach. The AUC variable will be analyzed by a t-test for unpaired data. A second analysis using a multivariate approach will be carried out for those factors considered as clinically relevant in relation to pain and therefore a logistic regression will be used.

Ethical Considerations: The study will be strictly conducted following the Declaration of Helsinki and the protocol and Standard Operating Procedures (SOPs) to ensure compliance with the Good Clinical Practice (GCP) standards. It is the responsibility of the researcher to obtain the valid informed consent from the guardian / legal representative, as the patient's condition will not allow to consent. Before obtaining the consent the investigator will explain to each guardian / legal representative the nature of the study, its purpose, the procedures, the estimated duration, the potential risks and benefits associated with the participation, as well as any inconvenience that this may involve.

Duration of Treatment: The treatment has a maximum duration of 60 min for each patient. The follow-up includes visits and has duration of 6 consecutive days.

Safety Assessment: Potential side effects of treatments will be recorded. Frequent adverse effects of fentanyl administration include respiratory depression, apnea, muscle rigidity, bradycardia and transient hypotension.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria:

1. Patients that will come with a minimum 24-hour schedule of mechanical ventilation (MV)
2. Patients men and women> 18 years and <85 years
3. Patients speak and / or understand the Castilian / Catalan
4. Patients with hemodynamic and respiratory stability enough, that allows mobilization procedure turn.
5. Patients who have a carer / guardian giving consent to participate in the study

Exclusion Criteria:

The subjects presenting one or more of the following criteria are NOT eligible to participate in this study:

1. Patients with known hypersensitivity to fentanyl and muscle relaxants
2. Patients who are receiving a neuromuscular blocking Neurocritical
3. Patients serious (TCE and / or other severe neurological injury (Glasgow <8), increased intracranial pressure, peripheral neuropathy, quadriplegia)
4. Patients with brain death or vegetative state
5. Patients who have received some extra supplement opioids (morphine, Fentanest) bolus within 4 hours prior to the study.
6. Collaboration in the 30 days prior to any study either experimental drugs or devices.
7. Patients that potentially present alterations in the ability to understand when they are aware to understand the purpose of the study and to give informed consent in writing.
8. Patients undergoing treatment with Monoamine Oxidase Inhibitors
9. Women who are pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in the incidence of pain at the beginning and end of rotation | Expected average of 5 minutes
  Participants will be evaluated at the beginning and the end of rotation, an expected average of 5 minutes. The evaluation of the change in the incidence of pain will be done calculating the mean between the beginning and the end of rotation.

SECONDARY OUTCOMES:
Area under the curve (AUC) of incidence of pain (BPS) during mobilizations with spin | Since the end of the turn until 30 minutes after

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Roche-Campo, MD PhD, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Gemma Robleda, Rn PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Robleda G, Roche-Campo F, Sendra MA, Navarro M, Castillo A, Rodriguez-Arias A, Juanes-Borrego E, Gich I, Urrutia G, Nicolas-Arfelis JM, Puntillo K, Mancebo J, Banos JE. Fentanyl as pre-emptive treatment of pain associated with turning mechanically ventilated patients: a randomized controlled feasibility study. Intensive Care Med. 2016 Feb;42(2):183-91. doi: 10.1007/s00134-015-4112-7. Epub 2015 Nov 10. PMID 26556618
- [Derived] Robleda G, Roche-Campo F, Urrutia G, Navarro M, Sendra MA, Castillo A, Rodriguez-Arias A, Juanes-Borrejo E, Gich I, Mancebo J, Banos JE. A randomized controlled trial of fentanyl in the pre-emptive treatment of pain associated with turning in patients under mechanical ventilation: research protocol. J Adv Nurs. 2015 Feb;71(2):441-50. doi: 10.1111/jan.12513. Epub 2014 Aug 28. PMID 25168967